CLINICAL TRIAL: NCT05808140
Title: Clinical Application of Indocyanine Green Fluorescence Imaging to Assist Identification of Nerve Roots in Endoscopic Spinal Surgery
Brief Title: Fluorescence Imaging With Indocyanine Green(ICG) in Endoscopic Spinal Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Yuanlong Xie, Principal Investigator, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Yuanlong Xie
Record Dates: First submitted 2023-03-16; First posted 2023-04-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Disc Herniation
Keywords: Disc Herniation; Endoscopy; Indocyanine green; Near-infrared fluorescence imaging; Spinal nerve roots
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Indocyanine Green; Optical Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (No Intervention): Standard endoscopic spinal surgery
- 0.5mg/kg ICG group (Experimental): The patients receive 0.5mg/kg ICG intravenous injection before surgery. The search for lumbar nerve roots is performed with the assistance of fluoroscopic endoscopic imaging equipment. And the procedure follows standard endoscopic spinal surgery procedures.
  Interventions: Drug: Indocyanine Green; Device: Fluorescence imaging
- 1mg/kg ICG group (Experimental): The patients receive 1mg/kg ICG intravenous injection before surgery. The search for lumbar nerve roots is performed with the assistance of fluoroscopic endoscopic imaging equipment. And the procedure follows standard endoscopic spinal surgery procedures.
  Interventions: Drug: Indocyanine Green; Device: Fluorescence imaging
- 2mg/kg ICG group (Experimental): The patients receive 2mg/kg ICG intravenous injection before surgery. The search for lumbar nerve roots is performed with the assistance of fluoroscopic endoscopic imaging equipment. And the procedure follows standard endoscopic spinal surgery procedures.
  Interventions: Drug: Indocyanine Green; Device: Fluorescence imaging

INTERVENTIONS:
Drug: Indocyanine Green — Preoperatively, a single dose of intravenous indocyanine green is administered
  Other Names: ICG
  Arms: 0.5mg/kg ICG group; 1mg/kg ICG group; 2mg/kg ICG group
Device: Fluorescence imaging — Use of a spinal endoscopic fluorescent imaging system to assist surgeons in identifying and protecting nerve roots intraoperatively
  Arms: 0.5mg/kg ICG group; 1mg/kg ICG group; 2mg/kg ICG group

SUMMARY:
In endoscopic spinal nerve root decompression surgery, the intraoperative nerve exploration is time-consuming and critical. According to statistics, the incidence of nerve root injury under spinal endoscope is 1.8-2.5%. Damage to nerve roots may lead to postoperative sensory retardation and motor weakness, thereby impairing the physical function of patients. A real-time auxiliary intraoperative nerve identification technology is necessary.

In this prospective, open-label, randomized, parallel controlled trial, 40 patients who undergo endoscopic spinal surgery are included. Subjects are randomly divided into control group and low, medium and high Indocyanine green(ICG) preoperative administration experimental group. Standard endoscopic spinal surgery is performed in the control group. Patients in the experimental group received an intravenous injection of ICG before surgery, and a standard endoscopic spinal surgery is performed with the use of a fluoroscopic endoscopic surgical imaging system to assist the surgeon in identifying and protecting the nerve roots.

The main objectives of this experiment are (i) to explore the safety and feasibility of ICG fluorescence imaging to assist in nerve root identification during endoscopic spinal surgery and (ii) the effectiveness of this technique for endoscopic search for nerve roots. The secondary objective is to explore the optimal ICG dosing regimen.

DETAILED DESCRIPTION:
With the accelerated pace of the global aging society, the prevalence of degenerative diseases is increasing. At present, spinal degenerative diseases caused by body degeneration have become the most common type. With the continuous deepening of the research on spinal degenerative diseases and the continuous development, update and promotion of minimally invasive surgery technology and instruments, minimally invasive surgery has attracted more and more attention of spine surgeons due to its advantages of rapid recovery, small trauma and fewer complications.

The core of endoscopic spinal surgery is nerve root decompression. The procedure is centered on the nerve roots, which can be damaged with the slightest carelessness. According to statistics, the incidence of nerve root injury under spinal endoscope is 1.8-2.5%. Most of the injuries include the stimulation and edema of the nerve root during the operation, which may lead to postoperative sensory retardation and motor weakness, which will damage the patient's physical function and reduce overall satisfaction. The intraoperative nerve exploration is time-consuming and critical, and the variability of the patient's nerve anatomy will also add difficulties to the operation. A real-time auxiliary intraoperative nerve identification technology is necessary.

With the progress of optical technology, fluorescent-guided surgery has shown considerable prospects in assisting in identifying nerves. Indocyanine green (ICG) is the only fluorophore approved by the US Food and Drug Administration (FDA) for intraoperative near-infrared imaging. It can emit near-infrared light after being irradiated by excitation light, which has the characteristics of high penetration depth, low spontaneous fluorescence and high sensitivity. At present, ICG near-infrared fluorescence imaging has been applied to tumor detection, lymphangiography and vascular perfusion evaluation. In recent years, more and more researchers have paid attention to the application value of ICG fluorescence imaging in neuroimaging. It has been applied to clinical research of thoracic sympathetic ganglion, facial nerve, phrenic nerve and pelvic nerve.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lumbar disc herniation based on symptoms and Imaging examination
* Patients undergo endoscopy spinal surgery for nerve root decompression
* Patients have no clear contraindications to surgery, and has the ability to understand and act and has informed consent, and can participate in all study follow-up voluntarily and signe a written informed consent form.

Exclusion Criteria:

* The patients have thyroid related diseases, including autonomous nodules
* Patients are allergic to iodine or shellfish
* Patients have ankylosing spondylitis, lumbar instability or bony spinal stenosis
* Patients have diabetes, vascular related diseases, or abnormal liver and kidney function
* Difficulty in tolerating anaesthesia
* Pregnant or lactating women
* Patients are unable to communicate or do not follow directions
* The investigators consider the patient unsuitable to participate in this study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-12-14 (Actual); Study Completion 2025-12-14 (Actual)

PRIMARY OUTCOMES:
Fluorescence imaging rate of nerve roots | Intraoperative
  Number of the nerve roots with fluorescent imaging in the experimental group/Total nerve roots in the experimental group×100%
Fluorescence signal ratio of nerve root to back fluorescence | Immediately postoperative
  Nerve root fluorescence intensity/Background fluorescence intensity
Time taken to find the nerve root endoscopically | Intraoperative
  Time from opening the ligamentum flavum to finding the nerve root in spinal endoscopic procedures

SECONDARY OUTCOMES:
ICG-related adverse reactions | Immediately after ICG administration to 30 min after administration
Visual analogue pain scale (Visual analogue scale, VAS) | 1 day before surgery, 1 day after surgery, 1 week after surgery, 1 month after surgery
  The VAS pain score uses the VAS scale, with end 0 being no pain, graded 1-4 being mild pain, 5-6 being moderate pain, 7-9 being severe pain, and end 10 being unbearable pain. The higher the score, the more severe the pain level.
Oswestry disability index（ODI） | 1 day before surgery, 1 day after surgery, 1 week after surgery, 1 month after surgery
  The ODI score is based on the Oswestry Disability Index questionnaire. The lowest score was 0% and the highest score was 100%, with higher scores indicating more severe functional impairment.
Surgical complications | Within 1 week after surgery
  Record any surgical complications that occurred in the patient within 1 week after surgery
Length of surgery | From the beginning to the end of the surgery
  Use a timer to record the length of the surgery (accurate to the minute)

CONTACTS AND LOCATIONS:
Overall Officials: Yuanlong Xie, M.D., Principal Investigator — Department of Spine Surgery and Musculoskeletal Tumor, Zhongnan Hospital of Wuhan University
Locations (1):
- Department of Spine Surgery and Musculoskeletal Tumor, Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

REFERENCES:
- [Background] Gokaslan ZL, Telfeian AE, Wang MY. Introduction: Endoscopic spine surgery. Neurosurg Focus. 2016 Feb;40(2):E1. doi: 10.3171/2015.11.FOCUS15597. No abstract available. PMID 26828878
- [Background] Fourney DR, Dettori JR, Norvell DC, Dekutoski MB. Does minimal access tubular assisted spine surgery increase or decrease complications in spinal decompression or fusion? Spine (Phila Pa 1976). 2010 Apr 20;35(9 Suppl):S57-65. doi: 10.1097/BRS.0b013e3181d82bb8. PMID 20407352
- [Background] Strakowski JA. Ultrasound-Guided Peripheral Nerve Procedures. Phys Med Rehabil Clin N Am. 2016 Aug;27(3):687-715. doi: 10.1016/j.pmr.2016.04.006. Epub 2016 Jun 6. PMID 27468673
- [Background] He K, Zhou J, Yang F, Chi C, Li H, Mao Y, Hui B, Wang K, Tian J, Wang J. Near-infrared Intraoperative Imaging of Thoracic Sympathetic Nerves: From Preclinical Study to Clinical Trial. Theranostics. 2018 Jan 1;8(2):304-313. doi: 10.7150/thno.22369. eCollection 2018. PMID 29290809
- [Background] Kanno K, Aiko K, Yanai S, Sawada M, Sakate S, Andou M. Clinical use of indocyanine green during nerve-sparing surgery for deep endometriosis. Fertil Steril. 2021 Jul;116(1):269-271. doi: 10.1016/j.fertnstert.2021.03.014. Epub 2021 Apr 8. PMID 33840452
- [Background] Chen SC, Wang MC, Wang WH, Lee CC, Yang TF, Lin CF, Wang JT, Liao CH, Chang CC, Chen MH, Shih YH, Hsu SP. Fluorescence-assisted visualization of facial nerve during mastoidectomy: A novel technique for preventing iatrogenic facial paralysis. Auris Nasus Larynx. 2015 Apr;42(2):113-8. doi: 10.1016/j.anl.2014.08.008. Epub 2014 Sep 6. PMID 25199746
- [Background] He K, Li P, Zhang Z, Liu J, Liu P, Gong S, Chi C, Liu P, Chen C, Tian J. Intraoperative near-infrared fluorescence imaging can identify pelvic nerves in patients with cervical cancer in real time during radical hysterectomy. Eur J Nucl Med Mol Imaging. 2022 Jul;49(8):2929-2937. doi: 10.1007/s00259-022-05686-z. Epub 2022 Mar 1. PMID 35230489